CLINICAL TRIAL: NCT05069298
Title: Effect of Milk Thistle Derivative Silibinin(A) as a Potential Anti-obesity Agent
Brief Title: Effect of Silibinin(A) as a Potential Anti-obesity Agent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Juan Jose Hernández Morante, Main researcher at Eating-related disorders research unit, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIO-HPC_1
Record Dates: First submitted 2021-05-29; First posted 2021-10-06 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Overweight and Obesity; Hypercholesterolemia; Hypertriglyceridemia
MeSH Terms: conditions — Overweight; Obesity; Hypercholesterolemia; Hypertriglyceridemia | interventions — Silybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION (Experimental): Silibinin (A) for three months, with an administration regimen of 3 oral doses of 300 mg per day, before each main meal.
  Interventions: Dietary Supplement: Silibinin A
- CONTROL (Placebo Comparator): Similar treatment regimen, but with a placebo.
  Interventions: Dietary Supplement: Silibinin A

INTERVENTIONS:
Dietary Supplement: Silibinin A — The compound will be administered following a 300 mg / 3 day schedule, before each main meal.
  Other Names: Milk thistle derivative

SUMMARY:
Our preliminary reports have found in silico and in vitro that the milk thistle derivative Silibinin(A) is able to inhibit pancreatic lipase, in a similar way that the classical anti-obesity drug orlistat.

Therefore, the investigators want to carry out the present trial in order to confirm that Silibinin(A) is able to in vivo inhibit pancreatic lipase, which will reduce the fat absorption and therefore will decrease the amount of energy from food intake.

Considering that milk thistle has been extensively studied in humans as liver-protector, the investigators consider that the use of human subjects will be of great interest to accelerate the employment of this compound to improve the effectiveness of dietary treatment in overweight/obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 24,9
* Voluntarily participate in the study

Exclusion Criteria:

* significant cognitive impairment
* psychiatric disorders
* chronic pharmacological treatment that may affect the effectiveness of the dietary intervention (corticosteroids, thyroid hormones, oral antidiabetic agents or lipid-lowering drugs)
* chronic disease that may interfere with dietary therapy (cancer, renal or hepatic impairment, chronic gastrointestinal conditions)
* acute disease episodes during the study
* subjects who followed a hypocaloric diet at the allocation time or in the 3 months prior to the beginning of the study
* pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-21 (Estimated)

PRIMARY OUTCOMES:
Percentage of total body weight loss | 3 months
  Change in body weight from baseline to the end of study period (3 months).

SECONDARY OUTCOMES:
Plasma total cholesterol | 3 months
  Change in plasma total cholesterol levels from baseline to the end of study period (3 months).
Plasma low density level cholesterol (cLDL) | 3 months
  Change in plasma cLDL levels from baseline to the end of study period (3 months).
Plasma triglycerides | 3 months
  Change in plasma triglyceride levels from baseline to the end of study period (3 months).
Body mass index (BMI) | 3 months
  Change in BMI from baseline to the end of study period.
Body fat percentage | 3 months
  Change in body fat from baseline to the end of study period.
Waist circumference | 3 months
  Change in waist circumference from baseline to the end of study period.

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Hernández Morante, PhD, Principal Investigator — Catholic University of Murcia
Locations (1):
- Faculty of Nursing. Catholic University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The data derived from the present trial will be located in public domain databases, concretely in the Mendeley data repository (https://data.mendeley.com/). Nevertheless, all data will be available by request to the main researcher, Dr. Juan José Hernández Morante (e-mail:jjhernandez@ucam.edu).

REFERENCES:
- See also: Webpage of the research group and contact info. — http://bio-hpc.ucam.edu/ucamhealth/
- See also: Webpage of other collaborators — http://bio-hpc.ucam.edu/